CLINICAL TRIAL: NCT06189742
Title: Tezepelumab in the Treatment of Co-morbid Allergic Rhinitis and Allergic Asthma Study (TEZARS) - An Open-Label Exploratory Mechanistic Pilot Study to Evaluate Tezepelumab Efficacy in Asthma and Allergic Rhinitis
Brief Title: Tezepelumab in Allergic Rhinitis and Asthma Study (TEZARS)
Acronym: TEZARS
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Anne Ellis (Other)
Responsible Party: Sponsor-Investigator, Dr. Anne Ellis, Professor, Department of Medicine, School of Medicine, and Department of Biomedical and Molecular Sciences, Queen's University; Director, Allergy Research Unit/Environmental Exposure Unit, Kingston Health Sciences Centre, KGH site, Queen's University
Organization: Queen's University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TEZARS-001
Record Dates: First submitted 2023-11-28; First posted 2024-01-03 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Asthma With Allergic Rhinitis
Keywords: Allergy; Allergic Rhinitis; Allergic Asthma; Allergic Asthma and Allergic Rhinitis; Tezepelumab; Seasonal allergies; Perennial allergies; Intermitent allergies; Persistant allergies
MeSH Terms: conditions — Hypersensitivity; Rhinitis, Allergic; Rhinitis, Allergic, Seasonal | interventions — tezepelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Non-allergic Participants (No Intervention)
- Allergic Participants (Experimental)
  Interventions: Biological: Tezepelumab

INTERVENTIONS:
Biological: Tezepelumab — Tezepelumab is a monoclonal antibody that blocks thymic stromal lymphopoietin (TSLP).
  Other Names: TEZSPIRE, tezepelumab-ekko
  Arms: Allergic Participants

SUMMARY:
The goal of this clinical trial is to learn about how well tezepelumab (pronounced TEZ e PEL ue mab), a Health Canada-approved drug for severe asthma, works in participants with coexisting allergic asthma and allergic rhinitis (hayfever). The main questions it aims to answer are:

* How well does the study drug work to reduce nasal symptoms following exposure to an allergen after 6 doses, and after 12 doses?
* Does the study drug reduce chemicals found in the nose known to be involved in the allergic rhinitis response?

Both allergic and non-allergic participants will be enrolled in the study.

Non-allergic participants will:

* Not be receiving the study drug.
* Be exposed to allergen via the Nasal Allergen Challenge, which involves the administration of allergen extract directly to the nose.
* Complete nasal symptom and quality of life questionnaires
* Have nasal fluid and blood samples collected at various time points up to 24 hours following allergen exposure.
* Visit the clinic 3 separate times:

  * At a screening visit to determine their eligibility to participate in the study
  * At the baseline Nasal Allergen Challenge visit
  * At the 24-hour post-Nasal Allergen Challenge follow-up visit

Allergic participants will:

* Receive one dose of tezepelumab every 1 month for 12 months. Tezepelumab will be administered as an injection into the fatty layer just beneath the skin on the stomach, arm, or thigh.
* Be exposed to allergen via the Nasal Allergen Challenge, which involves the administration of allergen extract directly to the nose.
* Complete nasal symptom and quality of life questionnaires
* Have nasal fluid and blood samples collected at various time points up to 24 hours following allergen exposure.
* Visit the clinic 17 separate times:

  * At a screening visit to determine their eligibility to participate in the study
  * At the baseline, 6-month, and 12-month Nasal Allergen Challenge visits
  * At each 24-hour post-Nasal Allergen Challenge follow-up visit
  * For each dose of the study drug

The investigator will compare changes in nasal symptoms and allergic chemicals measured from nasal fluid and blood samples between non-allergic participants and allergic participants at baseline and at 6- and 12-months following the use of the study drug.

DETAILED DESCRIPTION:
Tezepelumab is a novel monoclonal antibody that blocks thymic stromal lymphopoietin (TSLP), a molecule implicated in allergic disease. The purpose of this open-label, unblinded, exploratory mechanistic pilot study will be to evaluate the efficacy of tezepelumab (1 subcutaneous injection of 210mg given once every 4 weeks) in participants with moderate to severe allergic asthma and concomitant seasonal and perennial AR (SAR and/or PAR) over 12 months.

The tezepelumab in allergic rhinitis and asthma study (TEZARS) is a single-centre study. The trial will enrol 14 non-pregnant/non-lactating female and/or male comorbid allergic rhinitis (AR) and allergic asthma participants ages 18 to 65 years old from the Kingston, Frontenac, Lennox and Addington regions. An additional 5 non-allergic participants will be enrolled to participate in the baseline Nasal Allergen Challenge (NAC) visit and then will exit the study. Comorbid AR and allergic asthma participants attend the baseline NAC, then receive one dose of tezepelumab every 1 month for 12 months. A 6-month post-treatment follow-up NAC will be conducted one month following the sixth dose. A 12-month post-treatment follow-up NAC will be conducted two weeks following the twelfth dose. At each NAC visit, symptom scores and quality of life questionnaires, in addition to nasal fluid and blood samples will be collected at various time points.

The investigators hypothesize that tezepelumab will improve AR-related outcomes (TNSS; Peak Nasal Inspiratory Flow, PNIF; Rhinitis Control Assessment Test, RCAT) that are stimulated by NAC with seasonal and perennial allergens in our study population. Secondarily, the investigators hypothesize tezepelumab will decrease the release of allergic mediators (i.e., IL-1b, IL-3, IL-4, IL-5, IL-6, IL-8, IL-9 IL-10, IL-13, IL-18, MCP-1, TNFα, RANTES, eotaxin, tryptase, chymase) and alarmins (i.e., TSLP, IL-25, and IL-33) in the nose following NAC. A decrease in the gene expression of TSLP and mast cell mediators (tryptase and chymase) is also anticipated. Furthermore, the number of both nasal and peripheral eosinophils and total and specific immunoglobulin E (IgE) following NAC will decline after tezepelumab treatment. Five non-atopic controls will undergo baseline NAC to confirm the reliability of allergic mediator and alarmin methodologies. The investigators also hypothesize asthma-related outcomes (spirometry; Fractional Exhaled Nitric Oxide, FeNO; Asthma Control Questionnaire 5, ACQ5) will improve following treatment with tezepelumab. Finally, the NAC protocol in an asthmatic population will be assessed.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study, all participants should fulfil the following criteria based on local regulations:

1. Must be able and willing to provide written informed consent.
2. Must be willing and able to comply with the study requirements.
3. People between the ages of 18 and 65.
4. Body weight greater than 45 kg.
5. A person of childbearing potential must be either abstinent or using a medically acceptable method of birth control (see Section 3.5) and produce a negative urine pregnancy test at the screening visit and again at each treatment visit.

   For inclusion in the study, non-allergic participants should fulfil the following additional criteria based on local regulations:
6. Negative skin prick test to all relevant aeroallergen at screening with a wheal diameter no larger than that produced by the negative control.
7. Specific IgE levels to a relevant allergen are undetectable.
8. Negative screening Nasal Allergen Challenge, defined by a TNSS response of ≤ 3 (on a 12-point scale) and a decrease in PNIF of ≤ 30% after 10 minutes in response to a nasal application of a relevant aeroallergen extract.

   For inclusion in the study, allergic participants should fulfil the following additional criteria based on local regulations:
9. A minimum 2-year documented history of rhinoconjunctivitis symptoms to a relevant aeroallergen.
10. Positive skin prick test to a relevant aeroallergen at screening (matching the history in IC2) with a wheal diameter at least 5 mm larger than that produced by the negative control.
11. A minimum 2-year documented history of asthma, controlled with either moderate or high dose inhaled corticosteroids with or without another controller medication (long-acting beta-agonists and/or montelukast and/or a long-acting muscarinic antagonist.
12. Positive screening Nasal Allergen Challenge, defined by a TNSS response of ≥ 7 (on a 12-point scale) and a decrease in PNIF of ≥ 50% after 10 minutes in response to a nasal application of a relevant aeroallergen extract.

Exclusion Criteria:

Participants should not enter the study if any of the following exclusion criteria are fulfilled:

1. Involvement in the planning and/or conduct of the study (applies to both Investigator staff and/or staff at the study site).
2. Is unlikely to cooperate with the requirements of the study including having the ability to communicate with the investigator appropriately.
3. Inability to attend study visits or adhere to the study protocol, in the judgment of the principal investigator.
4. Previous enrolment in the present study.
5. Participation in another clinical study with an investigational product during the last 30 days.
6. Known hypersensitivity to the investigational product.
7. Currently uses or is expected to use any of the prohibited medications or other treatments as listed in Section 7.7.
8. An upper respiratory tract infection within 14 days of the NAC portion of the screening visit or baseline NAC visit.
9. History of immunological disorders or other diseases (including, but not limited to malignancy, cardiovascular, gastrointestinal, hepatic, renal, haematological, neurological, endocrine or pulmonary disease) that in the opinion of the investigator may pose additional risk factors for participation. Participants with basal cell carcinoma or squamous cell carcinoma that has been excised in the past 5 years may still participate in the study.
10. Nasal conditions that, according to the opinion of the investigator, may affect the outcome of the study, i.e. nasal septal perforation, current nasal polyps, other nasal malformations or history of frequent nosebleeds.
11. A known history of positive test results for Hepatitis B, Hepatitis C, HIV or tuberculosis other than what would be anticipated following vaccination.
12. Participant has a known history of current or previous parasitic infection.
13. Participant that is pregnant, lactating or actively trying to become pregnant.
14. Participant with a clinically relevant abnormality on physical examination.
15. Participant is unable to communicate or to understand the requirements of the study, which would impair communication between the participant and the investigator.
16. Significant history of alcohol or drug abuse, in the judgment of the investigator.
17. Serious asthma exacerbation requiring a hospital visit and/ or treatment with oral steroids within 4 weeks prior to screening.
18. FEV1 < 40 % predicted at screening.
19. Pre-NAC TNSS > 4 at the screening and baseline NAC visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Total Nasal Symptom Score (TNSS) | Baseline, 6 months, and 12 months
  To evaluate the effect of treatment with tezepelumab (210mg subcutaneous injection, once every 4 weeks for 12 doses) on TNSS (where a score of 0 indicates no nasal symptoms and 12 indicates the worst nasal symptoms) and 12 elicited by Nasal Allergen Challenge compared to baseline in a population with comorbid allergic rhinitis and allergic asthma.

SECONDARY OUTCOMES:
Peak Nasal Inspiratory Flow (PNIF) | Baseline, 6 months, and 12 months
  To evaluate the effect of treatment with tezepelumab (210mg subcutaneous injection, once every 4 weeks for 12 doses) on PNIF elicited by Nasal Allergen Challenge compared to baseline in a population with comorbid allergic rhinitis and allergic asthma.
Total Rhinoconjunctivitis Symptom Score (TRSS) | Baseline, 6 months, and 12 months
  To evaluate the effect of treatment with tezepelumab (210mg subcutaneous injection, once every 4 weeks for 12 doses) on TRSS (where a score of 0 indicates no rhinoconjunctivitis symptoms and a score of 24 indicates the most rhinoconjunctivitis symptoms) elicited by Nasal Allergen Challenge compared to baseline in a population with comorbid allergic rhinitis and allergic asthma.
Total Ocular Symptom Score (TOSS) | Baseline, 6 months, and 12 months
  To evaluate the effect of treatment with tezepelumab (210mg subcutaneous injection, once every 4 weeks for 12 doses) on TOSS (where a score of 0 indicates no ocular symptoms and a score of 9 indicates the most ocular symptoms) elicited by Nasal Allergen Challenge compared to baseline in a population with comorbid allergic rhinitis and allergic asthma.
Rhinitis Control Assessment Test (RCAT). | Each month for 12 months
  To evaluate the effect of treatment with tezepelumab (210mg subcutaneous injection, once every 4 weeks for 12 doses) on RCAT elicited by Nasal Allergen Challenge compared to baseline in a population with comorbid allergic rhinitis and allergic asthma. Six questions are ranked, and scores range between 1 (severely uncontrolled) and 5 (totally controlled).
Concentration of specific and total immunoglobulin E from nasal fluids. | Baseline, 6 months, and 12 months
  To evaluate the effect of treatment with tezepelumab on nasal and peripheral allergic biomarkers pre- and post-Nasal Allergen Challenge.
Concentration of tryptase from nasal fluids. | Baseline, 6 months, and 12 months
  To evaluate the effect of treatment with tezepelumab on nasal and peripheral allergic biomarkers pre- and post-Nasal Allergen Challenge.
Concentration of chymase from nasal fluids. | Baseline, 6 months, and 12 months
  To evaluate the effect of treatment with tezepelumab on nasal and peripheral allergic biomarkers pre- and post-Nasal Allergen Challenge.
Concentration of alarmins (TSLP, IL-33, IL-25) and type 2 cytokines (IL-4, Il-5, IL-13, etc.) from nasal fluids. | Baseline, 6 months, and 12 months
  To evaluate the effect of treatment with tezepelumab on nasal and peripheral allergic biomarkers pre- and post-Nasal Allergen Challenge.
Concentration of specific and total immunoglobulin E from serum. | Baseline, 6 months, and 12 months
  To evaluate the effect of treatment with tezepelumab on nasal and peripheral allergic biomarkers pre- and post-Nasal Allergen Challenge.
Concentration of tryptase from serum | Baseline, 6 months, and 12 months
  To evaluate the effect of treatment with tezepelumab on nasal and peripheral allergic biomarkers pre- and post-Nasal Allergen Challenge.
White blood cell count from whole blood. | Baseline, 6 months, and 12 months
  To evaluate the effect of treatment with tezepelumab on nasal and peripheral allergic biomarkers pre- and post-Nasal Allergen Challenge.
Forced Expiratory Volume for 1 second (FEV1) | Each month for 12 months
  To evaluate the effect of treatment with tezepelumab on asthma control following Nasal Allergen Challenge.
Peak Expiratory Flow Rate (PEFR) | Each month for 12 months
  To evaluate the effect of treatment with tezepelumab on asthma control following Nasal Allergen Challenge.
Fractional Exhaled Nitric Oxide (FeNO) | Baseline, 6 months, and 12 months
  To evaluate the effect of treatment with tezepelumab on asthma control following Nasal Allergen Challenge.
Asthma Control Questionnaire 5 (ACQ5). | Each month for 12 months
  To evaluate the effect of treatment with tezepelumab on asthma control following Nasal Allergen Challenge. Five questions are ranked, and scores range between 0 (totally controlled) and 6 (severely uncontrolled).

OTHER OUTCOMES:
Adverse reactions induced by Nasal Allergen Challenge | Baseline, 6 months, and 12 months
  To evaluate the safety of the current Nasal Allergen Challenge protocol in an asthmatic population through assessment of reported adverse events and required rescue medication.
Asthma symptoms induced by Nasal Allergen Challenge (symptom scores). | Baseline, 6 months, and 12 months
  To evaluate the safety of the current Nasal Allergen Challenge protocol in an asthmatic population based on symptom scores (ranked 0-3 including coughing, wheezing, chest tightness, shortness of breath).
Asthma symptoms induced by Nasal Allergen Challenge (spirometry). | Baseline, 6 months, and 12 months
  To evaluate the safety of the current Nasal Allergen Challenge protocol in an asthmatic population based on spirometry.

CONTACTS AND LOCATIONS:
Overall Officials: Anne K Ellis, MD, Principal Investigator — Queen's University
Locations (1):
- Kingston Health Sciences Centre- Kingston General Hospital, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No